CLINICAL TRIAL: NCT02087748
Title: A Randomized, Double-Blind, Within-Subject, Proof of Concept Study to Assess the Analgesic Efficacy and Safety of Voltaren Gel (1% Diclofenac Sodium) Compared to Placebo in Subjects Experiencing Delayed Onset Muscle Soreness
Brief Title: An Investigator Initiated, Within-Subject, Proof of Concept Study to Assess the Efficacy and Safety of Voltaren Gel in Subjects With DOMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lotus Clinical Research, LLC (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Neil Singla, Principal Investigator, Lotus Clinical Research, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCR-VOL-01C
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Pain; Delayed Onset Muscle Soreness
Keywords: DOMS
MeSH Terms: conditions — Pain | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1% diclofenac sodium gel (Active Comparator): Diclofenac sodium 1% gel 4 grams applied topically Q6 hour for 48 hours
  Interventions: Drug: 1% diclofenac sodium gel
- Placebo (Placebo Comparator): Placebo gel 4gm applied topically Q6 hour for 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1% diclofenac sodium gel — Diclofenac sodium 1% gel 4 grams applied topically Q6 hour for 48 hours
  Other Names: Voltaren
  Arms: 1% diclofenac sodium gel
Drug: Placebo — Placebo gel 4gm applied topically Q6 hour for 48 hours
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate analgesic efficacy of Topical Voltaren Gel (diclofenac sodium gel) 1% applied QID compared to Placebo in Subjects Experiencing Delayed Onset Muscle Soreness.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, placebo controlled, within-subject study is to evaluate the efficacy of topical diclofenac sodium gel (DSG) 1% in reducing pain associated with delayed onset muscle soreness (DOMS). Following exercise, subjects reporting significant DOMS received topical DSG 1% applied to 1 leg and placebo applied to the other every 6 hours for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide written informed consent prior to enrollment
* Male or female and 18 to 35 years of age.
* Patients who are not engaged in regular lower extremity fitness activities for more than 2 times per week for ≥2 consecutive weeks in the past 6 months prior to screening.
* Female patients are eligible only if all of the following apply:

  * Not pregnant (subjects of child bearing potential must have a negative beta human chorionic gonadotropin (β-hCG) pregnancy test at screening);
  * Not lactating;
  * Not planning to become pregnant within the duration of the study;
* Patients who are willing and capable of understanding and cooperating with the requirements of the study.
* Patients able to understand and communicate in English.

Randomization Inclusion Criteria:

* Patients who report a DOMS score ≥4 at rest (numerical rating scale of 0 to 10, where 0 is no pain and 10 is worst pain imaginable) secondary to delayed muscle soreness on both right and left legs. The DOMS scores at rest reported for each leg must be within 3 points of each other.
* Patients must report a categorical pain rating of moderate to severe for each leg on a scale of none, mild, moderate, or severe prior to randomization.

Exclusion Criteria:

* Have a body mass index of >32 kg/m2
* History of active or suspected esophageal, gastric, pyloric channel, or duodenal ulceration or bleeding within 30 days preceding screening.
* Psychiatric disease including major depression, bipolar disorder, or anxiety, or other medical condition that, in the opinion of the Investigator, would interfere with the evaluation of study drug efficacy or safety
* History of clinically significant cardiovascular, cerebrovascular, metabolic, pulmonary, neurological, hematological, autoimmune, psychiatric or endocrine disorders, including individuals with Type I or Type II diabetes, or other clinically significant medical condition that, in the opinion of the Investigator, may preclude safe study participation.
* Have had surgery or scheduled to undergo surgery of the hips or knees within 6 months prior to screening and/or during the study participation.
* Have significant biomechanical abnormality in the lower extremity that would preclude study evaluations, such as: peripheral or central neurological disease, significant back pain; symptomatic osteoarthritis of the hips, knew, or feet, or other painful conditions of the lower extremities.
* Have any type of orthopedic and/or prosthetic device or any skin abnormalities on the legs that may interfere with local tolerability.
* Currently taking corticosteroids or topical analgesic or anti inflammatory treatment whose the duration of action may affect study evaluations.
* Malignancy in the last 5 years, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin that has been surgically cured, or any Stage 1 cancer or carcinoma in situ cured by resection or localized radiation at least 5 years prior to screening with no evidence of recurrence.
* History of allergy (cutaneous or systemic), hypersensitivity, or asthma to any of the following: diclofenac, paracetamol, acetylsalicylic acid, salicylic acid, other NSAID or cyclooxygenase 2-specific inhibitor (COXIB) or known intolerance (cutaneous or systemic) to any of the ingredients in the gel, such as isopropyl alcohol or propylene glycol.
* History of known narcotic, analgesic, or alcohol abuse.
* Any cognitive impairment that would, in the opinion of the Investigator, preclude study participation or compliance with study procedures (e.g., Alzheimer's dementia).
* Previously received an investigational product within 30 days before the scheduled dose of study medication.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled in March 2014 and the last subject was enrolled in April 2014.
  Types of location: Investigative site was located at one research center.
Groups:
- 1% Diclofenac Sodium Gel: Diclofenac sodium 1% gel 4 grams applied topically Q6 hours for 48 hours to one leg, and placebo to the other leg.
Period: Overall Study
Arm/Group | 1% Diclofenac Sodium Gel
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One group will use 1% diclofenac sodium gel on the left leg and placebo on the right leg for the treatment duration. The other group will use the same products, but on opposite legs.
Arm/Group | 1% Diclofenac Sodium Gel
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (3.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in SPID Scores of DOMS on Walking Over 24 Hours
Description: The primary outcome is the analgesic efficacy of Topical Voltaren® gel compared to placebo in the reduction of the pain associated with DOMS. The statistical comparison of interest will be the mean reduction in DOMS scores upon walking in the leg receiving Topical Voltaren® gel vs the leg receiving placebo over the first 24 hours post treatment. Pain intensity was assessed at predefined time points (Predose, 3, 9, 15, 21, and 24 hours after first drug administration) using an 11-point Numeric Rating Scale (NPRS) where a score of zero indicates "no pain" and "10" indicates "pain as bad as you can imagine". Pain Intensity Differences at each predefined time point (calculated as post-baseline NPRS values - baseline NPRS values) were analyzed. The theoretical maximum range of Sum of pain intensity differences (SPID24) is from -50 (indicative of an increase in pain) to 50 (indicative of a decrease in pain).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1% Diclofenac Sodium Gel: Diclofenac sodium 1% gel 4 grams applied topically Q6 hours for 48 hours
  1% diclofenac sodium gel
- Placebo: Placebo gel 4gm applied topically Q6H for 48 hours
  Placebo: gel manufactured to mimic Diclofenac sodium1% gel
Arm/Group | 1% Diclofenac Sodium Gel | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 34.87 (22.86) | 23.62 (19.38)
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium Gel; Test type: Superiority or Other; p = 0.0324, t-test, 2 sided

2. Secondary Outcome: Mean Reduction in SPID Scores of DOMS at Rest Over 24 Hours
Description: The secondary outcome is the mean reduction in DOMS scores at rest in the leg receiving Topical Voltaren® gel versus the leg receiving placebo over the first 24 hours post treatment initiation.
  Pain intensity was assessed at predefined time points (at Predose, 3, 9, 15, 21, and 24 hours after first drug administration) using an 11-point Numeric Rating Scale (NPRS) where a score of zero indicates "no pain" and a score of 10 indicates "pain as bad as you can imagine". Pain Intensity Differences at each predefined time point (calculated as post-baseline NPRS values - baseline NPRS values) were analyzed. The theoretical maximum range of Sum of pain intensity differences (SPID24) is from -50 (indicative of an increase in pain) to 50 (indicative of a decrease in pain).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Diclofenac Sodium Gel | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 28.06 (23.84) | 24.81 (20.9)
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium Gel vs Placebo; Test type: Superiority or Other; p = 0.3688, t-test, 2 sided

3. Secondary Outcome: Mean Reduction in SPID Scores of DOMS While Standing Over 24 Hours
Description: The secondary outcome is the mean reduction in DOMS scores while standing in the leg receiving Topical Voltaren® gel versus the leg receiving placebo over the first 24 hours post treatment initiation.
  Pain intensity was assessed at predefined time points (at Predose, 3, 9, 15, 21, and 24 hours after first drug administration) using an 11-point Numeric Rating Scale (NPRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Pain Intensity Differences at each predefined time point (calculated as post-baseline NPRS values - baseline NPRS values) were analyzed. The theoretical maximum range of Sum of pain intensity differences (SPID24) is from -50 (indicative of an increase in pain) to 50 (indicative of a decrease in pain).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Diclofenac Sodium Gel | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 33.9 (23.29) | 21.62 (18.8)
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium Gel vs Placebo; Test type: Superiority or Other; p = 0.0275, t-test, 2 sided

ADVERSE EVENTS:
Description: For serious adverse events, events will be collected when identified from the date Subject signed Informed Consent up to 30 days after discontinuation from the study. For other adverse events, events will be collected until study completion or early termination.
Arm/Group | 1% Diclofenac Sodium Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No